CLINICAL TRIAL: NCT00893438
Title: Fatigue in Teenagers on the Internet (FitNet); Efficacy of Web-based Cognitive Behavioural Treatment for Adolescents With the Chronic Fatigue Syndrome
Brief Title: Efficacy of Web-based Cognitive Behavioural Treatment for Adolescents With Chronic Fatigue Syndrome
Acronym: FitNet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Innovatiefonds Zorgverzekeraars (Other)
Responsible Party: Principal Investigator, E.M. van de Putte, M.D. Ph.D., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZonMW-56100004; ISRCTN59878666
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome (CFS); Adolescence; Cognitive behaviour therapy (CBT); Web-based; Internet; Efficacy
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FitNet treatment (Experimental): FitNet treatment: web-based cognitive behaviour therapy
  Interventions: Behavioral: FitNet treatment
- Usual care (Active Comparator): waiting list for FitNet intervention (usual care allowed)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: FitNet treatment — web-based cognitive behavioural treatment for adolescents with CFS
  Other Names: CBT; Internet treatment
  Arms: FitNet treatment
Other: Usual care — Usual care treatment for adolescents with CFS
  Arms: Usual care

SUMMARY:
The aim of this study is to determine the efficacy of FITNET (web-based cognitive behavioural treatment) for adolescents with Chronic Fatigue Syndrome (CFS) in The Netherlands. The second goal of the study is to establish predictors of outcome. It is very important to know the characteristics of patients who will benefit from Cognitive Behavioural Treatment (CBT) and who will not. Possible predictors of outcome are: age, depression, anxiety, fatigue of the mother, parental bonding, self-efficacy, body consciousness of child and mother, physical activity (Actometer).

DETAILED DESCRIPTION:
All participants will be randomized to one of the two treatment arms:

1. Intervention with web-based cognitive behavioral treatment
2. Usual care

The duration of the cognitive behavioural program is limited to 6 months. The adolescents who have been assigned to the usual care will get the opportunity to attend the program after these 6 months. The total follow-up time is 12 months after the start of the web-based program.

The web-based program is developed for both the adolescents and the parents. The program consists of two parts, a psycho-educational part and a cognitive behavioural part consisting of 21 treatment modules. The therapist activates one or more treatment modules per week, dependent on the progress of the participant. Within a treatment module the participant will keep several journals, answer questions and do several assignments. All answers are sent to the therapist, with whom a weekly email contact will be realized.

Efficacy of the web-based program will be determined after 6 months. There will be a follow-up measurement at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (12 - 18 years) with Chronic Fatigue Syndrome

Exclusion Criteria:

* Score greater than or equal to 44 on the Stait-Trait Anxiety Inventory for Children
* Score greater than or equal to 20 on the Children's Depression Inventory
* No availability of computer and/or internet
* Risk of suicide
* Mental retardation

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
School presence | one year
Severity of fatigue | one year
Physical functioning as measured by the subscale physical functioning | one year

SECONDARY OUTCOMES:
Self-rated improvement | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sanne L Nijhof, MD, PhD-student, Principal Investigator — Wilhelmina Childrens' Hospital (University Medical Center Utrecht); Elise M van de Putte, MD, PhD, Study Director — Wilhelmina Childrens' Hospital (University Medical Center Utrecht); Gijs Bleijenberg, Prof, Study Director — University Medical Center St. Radboud; Cuno SP Uiterwaal, MD, PHD, Study Director — Julius Center for Health Sciences and Primary Care, University Medical Center Utrecht; Jan JL Kimpen, Prof., Study Director — UMC Utrecht
Locations (2):
- Netherlands (2):
  - University Medical Center St. Radboud, Nijmegen
  - Wilhelmina Childrens' Hospital (University Medical Center Utrecht), Utrecht

REFERENCES:
- [Derived] Collin SM, Nuevo R, van de Putte EM, Nijhof SL, Crawley E. Chronic fatigue syndrome (CFS) or myalgic encephalomyelitis (ME) is different in children compared to in adults: a study of UK and Dutch clinical cohorts. BMJ Open. 2015 Oct 28;5(10):e008830. doi: 10.1136/bmjopen-2015-008830. Erratum In: BMJ Open. 2019 Nov 20;9(11):e008830corr1. doi: 10.1136/bmjopen-2015-008830corr1. PMID 26510728
- [Derived] Nijhof SL, Bleijenberg G, Uiterwaal CS, Kimpen JL, van de Putte EM. Fatigue In Teenagers on the interNET--the FITNET Trial. A randomized clinical trial of web-based cognitive behavioural therapy for adolescents with chronic fatigue syndrome: study protocol. [ISRCTN59878666]. BMC Neurol. 2011 Feb 19;11:23. doi: 10.1186/1471-2377-11-23. PMID 21333021